CLINICAL TRIAL: NCT03804125
Title: A PHASE IV NON-INTERVENTIONAL STUDY. ADVERSE EVENTS (AES)/SUSPECTED ADVERSE DRUG REACTIONS (SADRS) ON THE PREVENTION OF STROKE AND SYSTEMIC EMBOLISM IN ADULT PATIENTS WITH NON-VALVULAR ATRIAL FIBRILLATION WITH ONE OR MORE RISK FACTORS AS PRIOR STOKE OR TRANSIENT ISCHAEMIC ATTACK; AGE >75; HYPERTENSION; DIABETES MELLITUS; SYMPTOMATIC HEART FAILURE (NYHA CLASS >II) AND PREVENTION OF VENOUS THROMBOEMBOLIC EVENTS (VTE) IN ADULT PATIENTS WHO HAVE UNDERGONE ELECTIVE HIP OR KNEE REPLACEMENT SURGERY UNDER TREATMENT WITH ELICUIS (REGISTERED) (APIXABAN)
Brief Title: A Study of Adverse Events and Suspected Adverse Drug Reactions in Patients Under Apixaban for Prevention of Stroke and Systemic Embolism With Non-Valvular Atrial Fibrillation and Venous Thromboembolic Events in Patients Who Have Undergone Elective Hip or Knee Replacement Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Company decision to not conduct the study and was cancelled prior to any enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661097; ELICUIS FV MEXICO (Other: Alias Study Number)
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Stroke; Thrombosis, Deep Vein; Pulmonary Embolism
MeSH Terms: conditions — Stroke; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months

SUMMARY:
To characterize and analyze the number, type and incidence of adverse events/suspected adverse drug reactions in patients treated with Apixaban, according to therapeutic indications approved in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Patients (men and women) over 18 years old.
* Patients who have received at least one dose of apixaban for prevention of stroke and systemic embolism with non-valvular atrial fibrillation with one or more of the following stroke risk factors: prior stoke or transient ischaemic attack; age >75; hypertension; diabetes mellitus; symptomatic heart failure (NYHA class >II); or for prevention of venous thromboembolic events (VTE) in adult patients who have undergone elective hip or knee replacement surgery.
* Subjects who are willing and able to comply with all scheduled visits.

Exclusion Criteria:

* Patients who have received apixaban in a clinical trial.
* Patients who received apixaban for another indication locally approved or have a contraindication according to the information to prescribe of the product in Mexico.
* Hypersensitivity to the active substance or to any of the excipients.
* Active clinically significant bleeding.
* Hepatic disease associated with coagulopathy and clinically relevant bleeding risk.
* Lesion or condition considered a significant risk factor for major bleeding. This may include current or recent gastrointestinal ulceration, presence of malignant neoplasms at high risk of bleeding, recent brain or spinal injury, recent brain, spinal or ophthalmic surgery, recent intracranial haemorrhage, known or suspected oesophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities.
* Concomitant treatment with any other anticoagulant agent e.g. unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin, etc.), heparin derivatives (fondaparinux, etc.), and oral anticoagulants (warfarin, rivaroxaban, dabigatran, etc.) except under specific circumstances of switching anticoagulant therapy. Concomitant medication with Nonsteroidal anti-inflammatory drugs (NSAIDs ).
* Pregnancy and breast-feeding.
* Severe acute or chronic psychiatric condition and other significant medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have received at least one dose of apixaban for prevention stroke and systemic embolism with non-valvular atrial fibrillation or for prevention of venous thromboembolic events (VTE) in adult patients who have undergone elective hip or knee replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
the number and type of suspected adverse drug reactions, including serious and non-serious cases | 48 months
  To characterize and to analyze the number, type and incidence of suspected adverse drug reaction (SADRs) in patients receiving apixaban according to the therapeutic indications approved in Mexico:
  A. Prevention of stroke and systemic embolism in adult patients with non-valvular atrial fibrillation with one or more risk factors as prior stoke or transient ischaemic attack; age >75; hypertension; diabetes mellitus; symptomatic heart failure (NYHA class >II) B. and in prevention of venous thromboembolic events (VTE) in adult patients who have undergone elective hip or knee replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.